CLINICAL TRIAL: NCT01146132
Title: Nutrition and Physical Activity in Patients With Cerebrovascular Disease
Acronym: ALVINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manon Gantenbein (Other)
Collaborators: Centre Hospitalier du Luxembourg (Other)
Responsible Party: Sponsor-Investigator, Manon Gantenbein, Clinical Research Coordinator, Public Research Centre Health, Luxembourg
Organization: Public Research Centre Health, Luxembourg (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CRP-Santé
Record Dates: First submitted 2010-06-15; First posted 2010-06-17 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Cerebrovascular Disorders
Keywords: Nutrition; Physical activity; Cerebrovascular disease; wine consumption; BMI; Pulse transit time; transcranial Doppler sonography
MeSH Terms: conditions — Cerebrovascular Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Luxembourg diet + wine (Other): Luxembourg variant of the mediterranean Diet, physical activity with wine consumption
  Interventions: Dietary Supplement: Luxembourg variant of Mediterranean diet + physical activity +/- wine
- conventional + wine (Other): conventional Diet with red wine
  Interventions: Dietary Supplement: Conventional diet +/- wine
- conventional (Other): conventional diet without wine
  Interventions: Dietary Supplement: Conventional diet +/- wine
- Luxembourg diet (Other): Luxembourg variant of the mediterranean Diet, physical activity with wine consumption
  Interventions: Dietary Supplement: Luxembourg variant of Mediterranean diet + physical activity +/- wine

INTERVENTIONS:
Dietary Supplement: Conventional diet +/- wine — usual eating habits
  Arms: conventional; conventional + wine
Dietary Supplement: Luxembourg variant of Mediterranean diet + physical activity +/- wine — Walnuts, almonds, mustard and soy bean products as part of the Indo-Mediterranean diet could be recommended to ensure a variety of food constellation, as well as dark chocolate. This form of diet will be addressed to as "Luxembourg variant of the Mediterranean diet"
  Arms: Luxembourg diet; Luxembourg diet + wine

SUMMARY:
The study will provide evidence of eating habits and physical activity in cerebrovascular patients in Luxembourg and of the degree to which these habits may be changed acutely (after one month) and in the long run (after 4 months) by intensive counselling. Furthermore the influence of intensive counselling and of the consumption of red wine on cerebrovascular risk factors, cognition, and on surrogate parameters for stroke will be assessed.

DETAILED DESCRIPTION:
Quality of life in the elderly and their families is severely affected by stroke and cognitive dysfunction caused by atherosclerosis of the brain supplying arteries. Nutrition, namely a Mediterranean-style diet, nuts, soybean products, whole grain products, dark chocolate, fish oil and avoidance of salt, and regular physical activity play a major role in the prevention of these diseases. Data are available on cardiac patients, however little is known on cerebrovascular patients. The role of red wine in the protection of cerebrovascular disease is discussed; it may be simply an epiphenomenon of otherwise healthy lifestyle in the population with a regularly low alcohol consumption not properly corrected for in epidemiological studies. No prospective randomised data is available.

We intend to perform a prospective randomised study on nutrition and physical activity in 100 patients with chronic cerebrovascular disease (i.e. patients with atherosclerotic stenosis, at least 20% of a brain supplying artery as demonstrated by carotid ultrasound and without an acute stroke/TIA). The study consists of three parts:

(1) Assessment of eating and physical activity habits in these patients and correlation with indicators of cerebrocardiovascular disease (cerebral perfusion as measured by transcranial Doppler sonography, pulsatility of the transcranial and extracranial Doppler signal, elasticity of the carotid artery, ankle-brachial index, cognitive functioning) and risk factors of cerebrovascular disease (blood pressure and blood pressure amplitude assessed by 24 h ambulatory blood pressure measurement; HDL, LDL, triglycerides, Lp(a), glucose, HbA1c, homocysteine, and fibrinogen; waist-hip ratio and BMI).

2) Half of these patients will be randomised to intensive counselling concerning healthy eating and physical activity habits during the first month once a week. All the 100 patients will be reassessed after one month and after 4 months with the above mentioned parameters.

3) In a double cross-over design half of the patients allocated to intensive counselling (i.e. n=25) and half of the patients without intensive counselling (n=25) will be allocated to 0,2 l of red wine daily (men) or 0,1l of red wine daily (women), respectively. The remaining 50 patients will be advised to avoid red wine for the time of the study.

ELIGIBILITY:
Inclusion Criteria:

* In- and outpatients of the Neurology Department of the CHL and their family members
* Carotid atherosclerosis assessed by B-mode ultrasound of at least 20% lumen reduction
* No acute stroke/TIA/amaurosis fugax (at least 3 months ago)
* Temporal ultrasound window suitable for recording of the middle cerebral artery
* Ability to give informed consent

Exclusion Criteria:

* No signed informed consent
* patient not able to give informed consent

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Differences in mean systolic blood pressure in the two diet/sport arms | 4 months
  Assess the influence of intensive counselling and of the consumption of red wine on cerebrovascular risk factors, cognition and on surrogate parameters for cerebrovascular disease.

SECONDARY OUTCOMES:
Effects on cerebrovascular health profile | 4 months
  Assess effects on cerebrocardiovascular health profile, cognitive function and ultrasound parameters.
Assessment of genetic marker and/or genetic modifications. | Baseline
  The genetic analyses will investigate:
  A) Profiles of inflammatory, anti-inflammatory cytokines B) Genes related to risk of stroke C) Chromosome regions related to atherosclerosis D) Genetic polymorphism in inflammation
  Genes to be analyzed: FABP2, MTP1, ApoE, ApoA1, PPAR gamma Pro 12 Ala, TNF alpha, Paraoxonase 1, ADH, Kinesin-like protein (KIF) 6 Trp719Arg (rs20455), SNP, 5 (component of complement 5) 2416A> G variant (rs17611), sCAMs (sICAM-1, sVCAM-1, sPSEL et sESEL), (C3, C4) Complement and CRP, P-selectin and its ligand, P-selectin glycoprotein ligand 1

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Droste, Pr, MD, Principal Investigator — Centre Hospitalier du Luxembourg
Locations (1):
- CHL, Luxembourg, Luxembourg

REFERENCES:
- [Derived] Droste DW, Iliescu C, Vaillant M, Gantenbein M, De Bremaeker N, Lieunard C, Velez T, Meyer M, Guth T, Kuemmerle A, Gilson G, Chioti A. A daily glass of red wine associated with lifestyle changes independently improves blood lipids in patients with carotid arteriosclerosis: results from a randomized controlled trial. Nutr J. 2013 Nov 15;12(1):147. doi: 10.1186/1475-2891-12-147. PMID 24228901